CLINICAL TRIAL: NCT01755858
Title: A Phase 2a, Placebo-controlled Trial to Evaluate the Impact of Intravenous Bendavia™ on Ischemia Reperfusion Injury in Atherosclerotic Renal Artery Stenosis in Patients Undergoing Percutaneous Transluminal Angioplasty of the Renal Artery
Brief Title: Effects of Intravenous Bendavia™ on Reperfusion Injury in Patients Undergoing Angioplasty of the Renal Artery
Acronym: EVOLVE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SPIRI-225
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Renal Artery Obstruction; Hypertension, Renovascular; Ischemia Reperfusion Injury
Keywords: elamipretide
MeSH Terms: conditions — Renal Artery Obstruction; Hypertension, Renovascular; Reperfusion Injury | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bendavia (Experimental): Bendavia, intravenous infusion, 0.05 mg/kg/hr for a maximum duration of 4 hours.
  Interventions: Drug: Bendavia
- Placebo (Placebo Comparator): Placebo (no active drug), intravenous infusion, for a maximum duration of 4 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bendavia
  Other Names: MTP-131; Elamipretide
  Arms: Bendavia
Drug: Placebo
  Arms: Placebo

SUMMARY:
This was a Phase 2a prospective, single center, randomized, double-blind, placebo-controlled study designed to assess the efficacy, pharmacokinetics, safety and tolerability of IV elamipretide for reduction of reperfusion injury in subjects with Atherosclerotic Renal Artery Stenosis (ARAS), who are undergoing percutaneous transluminal angioplasty of the renal artery (PTRA).

DETAILED DESCRIPTION:
This was a Phase 2a prospective, single center, randomized, double-blind, placebo-controlled study designed to assess the efficacy, pharmacokinetics, safety and tolerability of IV elamipretide for reduction of reperfusion injury in subjects with ARAS, who are undergoing percutaneous transluminal angioplasty of the renal artery (PTRA).

The randomization (1:1 active:placebo) was stratified by a diagnosis of diabetes mellitus. Participants received either 0.05 mg/kg/h elamipretide or matching placebo, administered as an IV infusion at 60 mL/h infused 30 minutes before and continued 3 hours after PTRA of the renal artery. After completion of the PTRA and stenting, subjects were to receive standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 and ≤80 years old.
* Patients with hypertension (systolic blood pressure [BP] >155 mm Hg) and/or requiring 2 or more antihypertensive medications: no restrictions will be placed on antihypertensive agents, although loop diuretics will be temporarily changed to diluting site agents (eg, hydrochlorothiazide, indapamide, metolazone) prior to each blood oxygen level-dependent magnetic resonance imaging (BOLD-MRI) study performed during the trial, unless, in the judgment of the Investigator, the change represents a hazard to the patient. ARAS patients will be identified based upon radiologic and clinical criteria suggestive of renovascular hypertension and/or hemodynamically significant renovascular disease >60% lumen occlusion (determined by quantitative computed tomography angiography or Doppler ultrasound velocity >200 cm/sec).
* Have an estimated glomerular filtration rate of ≥15 ml/min/1.73 m2 calculated using the Modification of Diet in Renal Disease (MDRD) formula.
* Have no contraindications to angiography such as severe contrast allergy.
* Have no contraindications to non-contrast magnetic resonance evaluations such as a pacemaker or magnetically active metal fragments.
* Able to comply with protocol.
* Women of childbearing age must:
* Have a negative pregnancy serum human chorionic gonadotropin test prior to receiving study drug.
* Agree to use two forms of contraception for 3 months following receipt of the study drug.
* Men who are sexually active and able to father a child, must agree to use one of the birth control methods listed below for the entire study and for at least 2 months after receiving the study drug:
* Barrier methods (such as a condom or diaphragm) used with a spermicide.
* Hormonal methods used by his partner, such as birth control pills, patches, injections, vaginal ring, or implants.
* Intrauterine device (IUD) used by his partner.
* Abstinence (no sex).
* Competent and able to provide written informed consent

Exclusion Criteria:

* Advanced chronic kidney disease defined as either Stage 5 or end-stage renal disease requiring dialysis.
* Have other clinically significant abnormalities or laboratory results that would, in the opinion of the investigators, compromise the safety of the patient including evidence of diabetic ketoacidosis, paraproteinemia, or triglycerides above 600 mg/dL.
* Clinically significant medical conditions within the six months before administration of Bendavia (e.g., cancer, stroke, myocardial infarction, active angina, congestive heart failure) that would, in the opinion of the investigators, compromise the safety of the patient.
* Have received an investigational drug within thirty (30) days of baseline.
* Have a serum sodium <135 mmol/L on the day of, and prior to, the PTRA.
* Are pregnant or breast feeding.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen C Textor, MD, Principal Investigator — Mayo Clinic; Richard Straube, MD, Study Director — Stealth BioTherapeutics Inc.
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Saad A, Herrmann SMS, Eirin A, Ferguson CM, Glockner JF, Bjarnason H, McKusick MA, Misra S, Lerman LO, Textor SC. Phase 2a Clinical Trial of Mitochondrial Protection (Elamipretide) During Stent Revascularization in Patients With Atherosclerotic Renal Artery Stenosis. Circ Cardiovasc Interv. 2017 Sep;10(9):e005487. doi: 10.1161/CIRCINTERVENTIONS.117.005487. PMID 28916603

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bendavia | Placebo
Started | 7 | 9
Completed | 6 | 8
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bendavia | Placebo | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (6.41) | 72.6 (7.78) | 69.8 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 3 | 6 | 9
Diabetes Mellitus Status [Count of Participants; unit: Participants]
  Positive | 0 | 3 | 3
  Negative | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Glomerular Filtration Rate (GFR), as Measured by Iothalamate Clearance, at Baseline (Pre-percutaneous Renal Artery Angioplasty and 8 Weeks Post-PTRA.
Description: Change in mean glomerular filtration rate (GFR), as measured by iothalamate clearance, from baseline (pre-percutaneous renal artery angioplasty, or pre-PTRA) and 8 weeks post-PTRA..
Time Frame: Baseline (pre-PTRA) and 8 weeks post-PTRA
Population: All participants for whom GFR by iothalamate clearance was measured at Baseline (pre-PTRA) and 8 weeks post-PTRA.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Bendavia | Placebo
Number analyzed (Participants) | 6 | 8
mL/min | 6.3 (12.14) | 12.0 (23.84)

2. Secondary Outcome: Change in Mean Glomerular Flow Rate as Measured Using Multi-Detector Computed Tomography (MDCT) at Baseline (Pre-PTRA) and 8 Weeks Post-PTRA.
Description: Change in mean glomerular flow rate as measured using Multi-Detector Computed Tomography (MDCT) at baseline (pre-PTRA) and 8 weeks post-PTRA, stented quantifiable scanned kidneys.
Time Frame: Baseline (pre-PTRA) and 8 weeks post-PTRA
Population: All participants with stented quantifiable kidneys for whom GFR by MDCT was measured at Baseline (pre-PTRA) and 8 weeks post-PTRA.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Bendavia | Placebo
Number analyzed (Participants) | 5 | 5
mL/min
  Right Single Kidney | 0.238 (0.2557) | 0.010 (0.0552)
  Left Single Kidney | 0.012 (0.1487) | 0.120 (0.1600)

3. Secondary Outcome: Change in Mean Regional Perfusion as Measured by MDCT at Baseline (Pre-PTRA) and 8 Weeks Post-PTRA
Description: Change in mean regional perfusion as measured by Multi-Detector Computed Tomography (MDCT) Baseline (pre-PTRA) and 8 weeks post-PTRA for stented quantifiable scanned kidneys.
Time Frame: Baseline (pre-PTRA) and 8 weeks post-PTRA
Population: All participants for whom regional perfusion was measured by MDCT with stented quantifiable scanned kidneys at Baseline (pre-PTRA) and 8 weeks post-PTRA.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Bendavia | Placebo
Number analyzed (Participants) | 5 | 5
mL/min
  Right Cortical | 1.266 (0.9341) | -0.816 (0.6614)
  Right Medullary | 0.242 (0.4143) | -0.082 (0.2541)
  Left Cortical | 0.614 (1.2390) | 0.220 (0.9112)
  Left Medullary | 0.150 (0.3788) | 0.156 (0.5184)

4. Secondary Outcome: Change in Mean Renal Blood Flow as Measured Using Multi-Detector Computed Tomography (MDCT) at Baseline (Pre-PTRA) and 8 Weeks Post-PTRA
Description: Change in mean renal blood flow (ml/minute) as measured using Multi-Detector Computed Tomography (MDCT) at Baseline (pre-PTRA) and 8 weeks post-PTRA for stented quantifiable scanned kidneys
Time Frame: Baseline (pre-PTRA) and 8 weeks post-PTRA
Population: All participants for whom renal blood flow as measured by MDCT was measured in stented quantifiable scanned kidneys at baseline and 8 weeks post-PTRA.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Bendavia | Placebo
Number analyzed (Participants) | 5 | 5
mL/min
  Right Cortical | 85.056 (63.2943) | -28.406 (54.8919)
  Right Medullary | 6.658 (20.3007) | -10.204 (21.2044)
  Right Total | 91.712 (82.4794) | -38.608 (43.4011)
  Left Cortical | 23.928 (64.4891) | 35.090 (59.9470)
  Left Medullary | 3.610 (14.4951) | 5.930 (19.0256)
  Left Total | 27.538 (78.0728) | 41.018 (75.6824)

5. Secondary Outcome: Change in Mean Renal Volume as Measured by Multi-Detector Computed Tomography (MDCT) at Baseline (Pre-PTRA) and 8 Weeks Post-PTRA.
Description: Change in mean renal volume as measured by Multi-Detector Computed Tomography (MDCT) at Baseline (pre-PTRA) and 8 weeks post-PTRA.
Time Frame: Baseline (Pre-PTRA) and 8 (+4) weeks post-PTRA
Population: All participants for whom renal volume was measured at baseline (Pre-PTRA) and 8 weeks post-PTRA in stented quantifiable kidneys.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Bendavia | Placebo
Number analyzed (Participants) | 5 | 5
mL
  Right Total Kidney Volume | 1.270 (12.8218) | 4.708 (13.7198)
  Left Total Kidney Volume | 5.090 (17.6951) | 10.220 (8.9447)
  Right Cortical | 4.372 (10.5438) | 9.840 (13.1156)
  Right Medullary | -3.162 (4.7616) | -5.132 (7.0670)
  Left Cortical | 4.534 (15.0459) | 10.100 (10.8462)
  Left Medullary | 0.558 (3.1016) | 0.120 (8.6277)

6. Secondary Outcome: Mean Change in Renal Oxygenation, Axial Aspect, in Stented Kidneys From Baseline (Pre-PTRA), and 27 Hours Post-PTRA and 8 Weeks Post-PTRA
Description: Mean change in renal oxygenation, axial aspect, in stented kidneys between baseline (pre-PTRA), and 27 hours post-PTRA and 8 weeks post-PTRA as measured by calculation of fractional hypoxia using blood oxygenation level-dependent magnetic resonance (BOLD-MR) imaging.
Time Frame: Baseline (Pre-PTRA) , 27 hours post-PTRA and 8 weeks post-PTRA
Population: All participants for whom fractional renal oxygenation, axial aspect, in stented kidneys was measured at baseline, 27 hours post-PTRA and 8 weeks post-PTRA.
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Bendavia | Placebo
Number analyzed (Participants) | 5 | 6
s^-1
  AxialRightPrefurosemideFractHyp%>20 27H Post PTRA | 13.440 (34.6825) | 16.708 (19.4980)
  AxialRightPrefurosemideFractHyp%>20; 8Wk Post PTRA: number analyzed (Participants) | 5 | 5
  AxialRightPrefurosemideFractHyp%>20; 8Wk Post PTRA | -3.380 (8.5013) | -10.892 (15.370)
  AxialRightPrefurosemideFractHyp%>30 27H PostPTRA | 5.206 (9.4875) | 11.600 (17.8192)
  AxialRightPrefurosemideFractHyp%>30 8Wk PostPTRA: number analyzed (Participants) | 5 | 5
  AxialRightPrefurosemideFractHyp%>30 8Wk PostPTRA | -2.120 (2.7426) | -1.840 (2.8693)
  AxialRightPostfurosemideFracHyp%>20 27HPostPTRA: number analyzed (Participants) | 5 | 5
  AxialRightPostfurosemideFracHyp%>20 27HPostPTRA | 24.280 (27.6206) | 13.854 (26.2292)
  AxialRightPostfurosemideFracHyp%>20 8WkPostPTRA: number analyzed (Participants) | 4 | 5
  AxialRightPostfurosemideFracHyp%>20 8WkPostPTRA | 28.625 (8.9537) | -7.560 (13.5471)
  AxialRightPostfurosemideFracHyp %30 27H Post PTRA: number analyzed (Participants) | 5 | 5
  AxialRightPostfurosemideFracHyp %30 27H Post PTRA | 6.080 (7.6904) | 13.490 (21.1322)
  AxialRightPostfurosemideFracHyp%>30 8WkPost PTRA: number analyzed (Participants) | 4 | 5
  AxialRightPostfurosemideFracHyp%>30 8WkPost PTRA | -0.400 (2.9473) | -1.370 (3.4412)
  AxialLeftPrefurosemide Frac Hyp%>20 27H Post PTRA | 1.320 (21.7694) | 12.767 (26.0745)
  AxialLeftPrefurosemide Frac Hyp%>20 8Wk Post PTRA: number analyzed (Participants) | 5 | 5
  AxialLeftPrefurosemide Frac Hyp%>20 8Wk Post PTRA | -0.420 (17.3066) | -8.160 (16.4477)
  AxialLeft Prefurosemide Frac Hyp %>30 27H PostPTRA | -3.128 (3.0154) | 16.938 (25.4089)
  AxialLeft PrefurosemideFrac Hyp %>30 8Wk PostPTRA: number analyzed (Participants) | 5 | 5
  AxialLeft PrefurosemideFrac Hyp %>30 8Wk PostPTRA | -0.602 (7.1510) | -6.360 (11.3054)
  AxialLeft Post-FurosemideFrac Hyp%>20 27HPostPTRA | 0.148 (21.0184) | 14.083 (34.6825)
  AxialLeft Post-FurosemideFrac Hyp%>20 8WkPostPTRA: number analyzed (Participants) | 5 | 5
  AxialLeft Post-FurosemideFrac Hyp%>20 8WkPostPTRA | -0.012 (17.3829) | -14.220 (13.303)
  AxialLeft Post-FurosemideFrac Hyp%>30 27HPostPTRA | -1.874 (2.5111) | 18.757 (27.1441)
  AxialLeft Post-FurosemideFrac Hyp%>30 8WkPostPTRA: number analyzed (Participants) | 5 | 5
  AxialLeft Post-FurosemideFrac Hyp%>30 8WkPostPTRA | 1.858 (7.0087) | -5.704 (8.3550)

7. Secondary Outcome: Mean Change in Renal Oxygenation, Coronal Aspect, in Stented Kidneys Between Baseline Pre-PTRA, 27 Hours Post-PTRA and 8 Weeks Post-PTRA
Description: Mean change in renal oxygenation, coronal aspect, in stented kidneys between baseline (pre-PTRA) and 27 hours post-PTRA or 8 weeks post-PTRA, as measured by calculation of fractional hypoxia using blood oxygenation level-dependent magnetic resonance (BOLD-MR) imaging, with and without Bendavia
Time Frame: 27H post PTRA and 8 weeks Post PTRA
Population: All participants for whom fractional renal oxygenation, coronal aspect, in stented kidneys was measured at baseline, 27 hours post-PTRA and 8 weeks post-PTRA.
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Bendavia | Placebo
Number analyzed (Participants) | 5 | 6
s^-1
  CoronalRtFractHypoxia% >20Prefuros.27HPost-PTRA | 20.314 (33.3525) | 9.083 (17.3368)
  CoronalRtFractHypoxia% >20Prefuros.8WkPost-PTRA: number analyzed (Participants) | 5 | 5
  CoronalRtFractHypoxia% >20Prefuros.8WkPost-PTRA | 4.140 (16.4690) | -2.220 (7.5549)
  CoronalRtFractHypoxia% >30Prefuros.27HPost-PTRA | 10.800 (9.6734) | 9.250 (30.6001)
  CoronalRtFractHypoxia% >30Prefuros8WkPost-PTRA: number analyzed (Participants) | 5 | 5
  CoronalRtFractHypoxia% >30Prefuros8WkPost-PTRA | 3.300 (10.1403) | -2.852 (11.1986)
  CoronalRtFractHypoxia% >20Postfuros27HPost-PTRA: number analyzed (Participants) | 4 | 5
  CoronalRtFractHypoxia% >20Postfuros27HPost-PTRA | 29.800 (33.5328) | 3.840 (22.4825)
  CoronalRtFractHypoxia% >20Postfuros8WKPost-PTRA: number analyzed (Participants) | 3 | 5
  CoronalRtFractHypoxia% >20Postfuros8WKPost-PTRA | 5.233 (7.5142) | -5.220 (4.6018)
  CoronalRtFractHypoxia% >30Postfuros27HPost-PTRA: number analyzed (Participants) | 4 | 5
  CoronalRtFractHypoxia% >30Postfuros27HPost-PTRA | 12.875 (13.2666) | 11.458 (32.8826)
  CoronalRtFractHypoxia% >30Postfuros8WkPost-PTRA: number analyzed (Participants) | 3 | 5
  CoronalRtFractHypoxia% >30Postfuros8WkPost-PTRA | 2.233 (3.5119) | -8.158 (16.5393)
  CoronalLeftFractHypoxia% >20Prefuros.27HPost-PTRA | 5.000 (23.7674) | 6.033 (31.1820)
  CoronalLeftFractHypoxia% >20Prefuros.8WkPost-PTRA: number analyzed (Participants) | 4 | 4
  CoronalLeftFractHypoxia% >20Prefuros.8WkPost-PTRA | -3.125 (10.2970) | -0.525 (12.5077)
  CoronalLeftFractHypoxia% >30Prefuros.27HPost-PTRA | -2.000 (8.9272) | 22.615 (35.6971)
  CoronalLeftFractHypoxia% >30Prefuros.8WkPost-PTRA: number analyzed (Participants) | 4 | 4
  CoronalLeftFractHypoxia% >30Prefuros.8WkPost-PTRA | -2.275 (4.4650) | -1.525 (12.3605)
  CoronalLeftFractHypoxia% >20Postfuros.27HPost-PTRA | 6.240 (24.5671) | 6.783 (29.1337)
  CoronalLeftFractHypoxia% >20Postfuros.8WkPost-PTRA: number analyzed (Participants) | 4 | 4
  CoronalLeftFractHypoxia% >20Postfuros.8WkPost-PTRA | 3.375 (9.2525) | -0.700 (14.7384)
  CoronalLeftFractHypoxia% >30Postfuros.27HPost-PTRA | 0.080 (7.3145) | 20.345 (31.5024)
  CoronalLeftFractHypoxia% >30Postfuros.8WkPost-PTRA: number analyzed (Participants) | 4 | 4
  CoronalLeftFractHypoxia% >30Postfuros.8WkPost-PTRA | -0.250 (2.0873) | -4.225 (12.7899)

8. Secondary Outcome: Mean Change in Systolic Blood Pressure Values (mmHg) From Pre-PTRA, Immediately Post-PTRA, 27 Hours and 8 (+4) Weeks Post-PTRA
Time Frame: Pre-PTRA and 27 hours post-PTRA and 8 weeks post-PTRA
Population: All participants for whom systolic blood pressure was measured at baseline (pre-PTRA) and 27 hours post-PTRA, or 8(+4) weeks post-PTRA.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Bendavia: Bendavia, intravenous infusion, 0.05 mg/kg/hr for a maximum duration of 4 hours.
  Bendavia
- Placebo: Placebo (no active drug), intravenous infusion, for a maximum duration of 4 hours.
  Placebo
Arm/Group | Bendavia | Placebo
Number analyzed (Participants) | 7 | 9
mmHg
  27 Hours Post-PTRA | -2.9 (14.78) | -3.8 (15.69)
  8 weeks Post PTRA: number analyzed (Participants) | 6 | 8
  8 weeks Post PTRA | 13.2 (19.88) | -0.8 (30.83)

9. Secondary Outcome: Mean Change in Diastolic Blood Pressure
Description: Mean Change in Diastolic Blood Pressure (DBP) values (mmHg) from baseline (pre-PTRA), immediately post-PTRA, 27 hours and 8 weeks post-PTRA, with and without Bendavia.
Time Frame: Pre-PTRA, immediately post-PTRA, 27 hours post-PTRA and 8 weeks post-PTRA
Population: All participants for whom diastolic blood pressure was measured.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bendavia | Placebo
Number analyzed (Participants) | 7 | 9
mmHg
  27 Hours Post-PTRA | 3.6 (7.76) | -2.0 (9.88)
  8 Weeks Post PTRA: number analyzed (Participants) | 6 | 8
  8 Weeks Post PTRA | 0.0 (9.70) | 0.1 (9.80)

ADVERSE EVENTS:
Arm/Group | Bendavia | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/9
Other Adverse Events (participants affected / at risk) | 2/7 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendavia (N=7) | Placebo (N=9)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bendavia (N=7) | Placebo (N=9)
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 1
Labile Blood Pressure (Vascular disorders) | 0 | 1
Blood sodium decreased (Investigations) | 1 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Pedal pulse decreased (Investigations) | 0 | 1
Thyroid function test abnormal (Investigations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less